CLINICAL TRIAL: NCT02385981
Title: Clinical Study to Review the Effects of an Auricular and Percutaneous Electric Stimulation of Nervus Vagus on the Oxygen Supply of Skin of Patients With Severe Claudicatio Intermittens
Brief Title: Vagal-stimulation-PAVK-tcpO2-study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Payrits, Thomas, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ASOKLIF 1301/PA
Record Dates: First submitted 2014-04-23; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Improvement of Skin Oxygen Supply

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stivax (Experimental): an intermittent stimulation of afferent vagus nerve at earlap
  Interventions: Device: Stivax

INTERVENTIONS:
Device: Stivax

SUMMARY:
H-1: tcpO2U2 > tcpO2U1 H-0: tcpO2U2 ≤ tcpO2U1

ELIGIBILITY:
Inclusion Criteria:

1. Each subject must sign an informed consent (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study.
2. PAVK stadium IIb due to Fontaine for at least 6 month
3. reduced systolic occlusion pressure at ankle (arteria tibialis posterior and anterior): ABI <0,9
4. radiologic significant occlusion at arteria femoralis superficialis and/or at arteria poplitea and/or at arteria of lower legs (MRT, CT, CO2-angiography or color-coded duplex sonography)
5. expected availability during study participation over 12 weeks (via health care center)

Exclusion Criteria:

1) <18 years 2) pregnancy and non-exclusion of pregnancy (women of child-bearing potential)

* 3)risk of incidence of pregnancy during study participation (female must fulfill one of the following criteria: menopause for more than 2 years, postmenopausal sterilisation, surgical sterilisation, hormonal contrazeption during study participation, spiral or diaphragm/condome+spermicide).

  4) lactation period 5) person of legal incapacity 6) regard, placement or appointment of an solicitor 7) military service 8) contraindication for the application of STIVAX 8a) malignant tumour (existence of a known, histologic verified, malignant tumour) 8b) hemophilia 8c) psoriasis vulgaris 8d) recent stroke 8e) superficial and deep infection of auricle and external auditory canal 9) (with the exception of STIVAX-application): foreseeable relevant stimulation of afferent contents of vagus to the ear within next 2 weeks.

  10) isolated diabetic microangiopathia 11) implantated cardiac pacemaker or defibrillator 12) transcutaneous partial pressure of oxygen (tcpO2) > 50 mmHg 13) concomitant disease with potential to limit the significance of the investigation of the walk distance (angina pectoris, heart failure, relevant pulmonary disease, relevant orthopedic or neurologic disease) 14) concomitant disease with potential to improve or to worsen the walking or the perfusion of the extremities in a relevant way.

  15) foreseeable change of PAVK-relevant medication or of concomitant medication with the potential to improve or to worsen the walking or the perfusion of the extremities in a relevant way within next 2 weeks.

  16) foreseeable start of a structured walking training within the next 2 weeks. 17) change in PAVK relevant medication or concomitant medication with potential to improve or worsen the walking or the perfusion of the extremities in a relevant way within the last 3 months.

  18) start with structured walking training within the last 3 months. 19) change in smoking habits within the last 3 months. 20) simultaneous participation in another clinical trial with insurance-protection.

  21) use of a therapy with stimulation of the afferent parts of vagus on the ear in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
change in transcutaneous oxygen partial pressure | 2015

SECONDARY OUTCOMES:
changes in SF 36 | 2015

OTHER OUTCOMES:
changes in ambulatory ability | 2015

CONTACTS AND LOCATIONS:
Locations (1):
- Landesklinikum Wiener Neustadt, Wiener Neustadt, Lower Austria, Austria